CLINICAL TRIAL: NCT01105728
Title: Endoscopic Resection of Gastric Subepithelial Masses, EndoResect Study
Acronym: EndoResect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Prof. Dr. Alexander Meining, Klinikum rechts der Isar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2632/09
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Gastric Subepitelial Mass
Keywords: Gastric subepitelial mass; Endoscopic full thickness resection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): Endoscopic resection
  Interventions: Procedure: Endoscopic resection

INTERVENTIONS:
Procedure: Endoscopic resection — Endoscopic resection of the gastric subepithelial mass

SUMMARY:
Gastric subepithelial masses might harbour gastrointestinal stromal tumors, which should get resected because of their malignant potential. To minimize the associated surgical trauma endoscopic endoluminal resection is favorable. Therefore in the current study endoscopic resection of gastric subepithelial masses is investigated. Since there is a certain risk of perforation due to the procedure, perforations get closed by placement of endoscopic clips (over-the-scope-clip [OTSC] clips).

DETAILED DESCRIPTION:
During an initial pilot phase 8 patients receive endoscopic resection under laparoscopic control. Thereafter and after positive initial results sole endoluminal endoscopy is done for a total of 38 patients.

ELIGIBILITY:
Inclusion Criteria:

* Endosonographically suspicous gastric subepithelial mass <=3 cm.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classes IV or V
* Pregnancy
* Bleeding disorders
* Contraindications for endoscopy
* Endosonographically shown large vessels in the area for resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
R0 Resection | 30 minutes
  Rate of R0 resections by an endoscopic approach for resection.

SECONDARY OUTCOMES:
Safety | 30 minutes
  Rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, MD, Principal Investigator — Klinikum rechts der Isar; Stefan von Delius, MD, Principal Investigator — Klinikum rechts der Isar; Hubertus Feußner, MD, Principal Investigator — Klinikum rechts der Isar; Dirk Wilhelm, MD, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany